CLINICAL TRIAL: NCT06818149
Title: A Study on the Clinical Classification and Outcome-Related Biological Markers of Immune Checkpoint Inhibitor-Related Myocarditis in Lung Cancer Patients
Brief Title: Biomarkers for Clinical Classification and Outcomes of Immune Checkpoint Inhibitor-Related-Related Myocarditis in Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Yanbin Kuang, Attending Physician,PhD, Shanghai Chest Hospital
Other Study IDs: IS24178
Record Dates: First submitted 2025-01-09; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer; Myocarditis Due to Drug
Keywords: Lung Cancer; Myocarditis; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Lung Neoplasms; Myocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Severe/critical group: Severe Type:
  Significant symptoms (e.g., fatigue, palpitations, chest pain) triggered by daily activities without hemodynamic changes; elevated myocardial biomarkers (Cardiac troponin, creatine kinase, Creatine kinase myocardial band, Aspartate aminotransferase，natriuretic peptides); new ECG changes; structural and functional myocardial abnormalities on echocardiography or MRI.
  Critical Type:
  Intolerable symptoms (e.g., respiratory dysfunction, heart failure, cardiogenic shock) at rest or minimal activity, with hemodynamic instability; significantly elevated myocardial biomarkers (Cardiac troponin, creatine kinase, Creatine kinase myocardial band, Aspartate aminotransferase, natriuretic peptides); severe myocardial structural and functional abnormalities on echocardiography or MRI; new severe arrhythmias on ECG .
  Interventions: Diagnostic Test: Biomarker Analysis for Severity Assessment
- Subclinical myocardial injury/mild group: Subclinical Myocardial Injury: All three of the following criteria must be met:
  1. No clinical symptoms triggered by daily activities;
  2. Only mild elevation of Cardiac troponin levels without elevation of other myocardial injury biomarkers;
  3. No abnormalities detected in other auxiliary examinations.
  Mild Type: The following conditions must be met for diagnosis:
  1. Daily activities may cause mild, nonspecific symptoms such as fatigue or shortness of breath;
  2. Mild elevation of myocardial injury biomarkers (Cardiac troponin, creatine kinase, Creatine kinase myocardial band, Aspartate aminotransferase，natriuretic peptides);
  3. Mild abnormalities on ECG, including new-onset sinus tachycardia, atrial arrhythmias, or nonspecific ST-T changes;
  4. No structural or functional abnormalities of the myocardium detected by echocardiography or cardiac MRI.
  Interventions: Diagnostic Test: Biomarker Analysis for Severity Assessment

INTERVENTIONS:
Diagnostic Test: Biomarker Analysis for Severity Assessment — Blood samples will be collected at baseline and at follow-up time points (3 days, 7 days, and before discharge). Traditional myocardial injury biomarkers, iron metabolism-related biomarkers, and immunological biomarkers will be tested.

SUMMARY:
This study aims to investigate the clinical classification and outcome-related biomarkers of immune checkpoint inhibitor (ICI)-related myocarditis in patients with lung cancer.A total of 50 patients with ICI-related myocarditis will be enrolled, including 25 with severe/critical myocarditis and 25 with subclinical/mild myocarditis. Blood samples will be collected at baseline and at follow-up time points (3 days, 7 days, and before discharge). Traditional myocardial injury markers, iron metabolism-related markers, and immunological markers will be measured and compared between groups. Changes in biomarkers after treatment will also be assessed. Clinical information such as in-hospital mortality and 3-month survival rates will be integrated to develop a severity assessment model. This model aims to evaluate disease severity and prognostic risk accurately by combining biomarkers, enhancing their application in clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed lung cancer and having received at least one dose of immune checkpoint inhibitor therapy;
* Clinically diagnosed with immune checkpoint inhibitor-related myocarditis;
* Aged 18 years or older;
* Voluntarily signed informed consent after being fully informed.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Presence of severe underlying cardiovascular diseases or recent acute cardiac events (e.g., myocardial infarction, severe arrhythmia);
* Concurrent other malignancies, immunosuppressive diseases, or autoimmune diseases;
* Inability to complete the required examinations and follow-ups specified in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with pathologically confirmed lung cancer who have received at least one dose of immune checkpoint inhibitor (ICI) therapy and have been clinically diagnosed with ICI-related myocarditis. Eligible participants must be 18 years or older and capable of providing informed consent. Patients will be stratified into two groups based on disease severity: severe/critical myocarditis and mild/subclinical myocardial injury. Exclusion criteria include pregnancy or breastfeeding, severe underlying cardiovascular diseases or recent acute cardiac events, concurrent other malignancies or immune-related diseases, and inability to complete required examinations and follow-ups. This population is intended to represent a clinically relevant cohort for exploring the association between biomarker dynamics and disease severity in ICI-related myocarditis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
The correlation between the dynamic changes in biomarker combinations and disease severity. | Up to 3 months
  By monitoring the dynamic changes in biomarker combinations at different time points (baseline, day 3, day 7, and before discharge), this study aims to evaluate the differences between the severe/critical group and the mild/subclinical myocardial injury group, and investigate their correlation with disease severity. Independent sample t-tests will be used to assess the differences between the two groups, assuming a moderate effect size (Cohen's d = 0.7) for biomarkers between the severe/critical and subclinical/mild immune checkpoint inhibitor-related myocarditis patients. If significant differences (p < 0.10) in biomarkers are observed between the groups, these differences will serve as key indicators for stratified management of disease severity.
Predictive performance of the severity assessment model | Up to 3 months
  The severity assessment model, constructed based on biomarker combinations, was evaluated for its predictive performance using indicators such as the ROC curve and AUC value. The model demonstrated a predictive performance with an AUC > 0.75 at different time points, indicating a high predictive ability and validating its practical application in clinical risk stratification.

SECONDARY OUTCOMES:
In-hospital mortality | Up to 3 months
  The rate of death occurring within the hospital during a patient's stay.
3-month survival rate | Up to 3 months
  The 3-month survival rate will be defined as the proportion of patients alive 3 months after enrollment in the study.
Improvement in patients' symptoms. | Up to 3 months
  Patients' symptom improvement (e.g., fatigue, dyspnea) will be recorded using the New York Heart Association (NYHA) Functional Classification and analyzed in relation to changes in biomarker combinations. This will provide insights into the potential application of biomarkers in predicting symptom improvement and disease severity.
Length of hospital stay. | Up to 3 months
  The length of hospital stay will be recorded and analyzed in relation to biomarker combinations and model prediction results, providing additional data to support practical applications in clinical management.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China